CLINICAL TRIAL: NCT02397824
Title: Orodental Manifestations of Rare Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: DC-2012-1677
Record Dates: First submitted 2015-03-11; First posted 2015-03-25 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Rare Disease Orodontal
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Salivary and blood samples

SUMMARY:
OroDental anomalies are one of the phenotypical aspects of at least 900 rare diseases or syndromes affecting by definition less than 1 in 2000 individual within the population (almost 25 million persons in Europe).

They are often described in association with other organs or system malformations, which is understandable, because the same genes and signalling pathways regulate the oral cavity formation or odontogenesis and the development of other organs. The various dental and orofacial anomalies can be classified by type (anomalies of tooth number, shape, size, structures of mineralized tissues, eruption, resorption, tumors; anomalies of oral mucosa; anomalies of tongue…), by signalling pathways and by syndrome families.

These anomalies (for example hypodontia/oligodontia, amelogenesis imperfecta, dentinogenesis imperfecta…) become increasingly identified as diagnostic and predictive traits. Not only is it important to recognise, name appropriately and integrate these dysmorphic clues into the patient dysmorphology analysis but it is essential to synthesize the observations and confront them to existing data about similar orodental anomalies encountered in some of the corresponding mutant mouse models.

Translational approaches in development and medicine, are relevant to gain understanding of molecular events underlying clinical manifestations and to enhance diagnostic accuracy.

The aim of this study is to improve the knowledge, diagnosis and care of oral cavity pathologies encountered in rare diseases via the identification and gathering of national and international patient cohorts and to structure the molecular diagnosis behind these conditions via targeted next-generation sequencing assays. Data collection is implemented on validated accredited tools (databases) complying with the legal regulations about patient data protection and medical record collection. All information is anonymized.

New effective diagnosis and therapeutic tools are being developed.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with a rare disease

  * New patient or patient already known in the center
  * Child (in his primary dentition) or adult
  * Man or woman
  * Having signed a consent form or accepted to participate to the study
  * Patient affiliated to social security
  * Validation of the inclusion by the principal investigator looking at the patient file

Exclusion Criteria:

* Patient whose clinical diagnostic is not possible

  * Patient whose clinical file does not contain teeth photos
  * Patient who has not signed a consent form and accepted to participate to the study
  * Patient who is not affiliated to social security.
  * Non validation of the inclusion by the principal investigator looking at the patient file

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Routine care hospitalization patient
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Dental history | baseline
  enamel defect
Familial history | baseline
  dental defect in family's subject
Familial genotyping | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- BLOCH-ZUPAN Agnès, Strasbourg, Alsace, France

REFERENCES:
- [Result] Gasse B, Prasad M, Delgado S, Huckert M, Kawczynski M, Garret-Bernardin A, Lopez-Cazaux S, Bailleul-Forestier I, Maniere MC, Stoetzel C, Bloch-Zupan A, Sire JY. Evolutionary Analysis Predicts Sensitive Positions of MMP20 and Validates Newly- and Previously-Identified MMP20 Mutations Causing Amelogenesis Imperfecta. Front Physiol. 2017 Jun 14;8:398. doi: 10.3389/fphys.2017.00398. eCollection 2017. PMID 28659819
- [Result] Rey T, Tarabeux J, Gerard B, Delbarre M, Le Bechec A, Stoetzel C, Prasad M, Laugel-Haushalter V, Kawczynski M, Muller J, Chelly J, Dollfus H, Maniere MC, Bloch-Zupan A. Protocol GenoDENT: Implementation of a New NGS Panel for Molecular Diagnosis of Genetic Disorders with Orodental Involvement. Methods Mol Biol. 2019;1922:407-452. doi: 10.1007/978-1-4939-9012-2_36. PMID 30838594
- [Result] Laugel-Haushalter V, Bar S, Schaefer E, Stoetzel C, Geoffroy V, Alembik Y, Kharouf N, Huckert M, Hamm P, Hemmerle J, Maniere MC, Friant S, Dollfus H, Bloch-Zupan A. A New SLC10A7 Homozygous Missense Mutation Responsible for a Milder Phenotype of Skeletal Dysplasia With Amelogenesis Imperfecta. Front Genet. 2019 May 28;10:504. doi: 10.3389/fgene.2019.00504. eCollection 2019. PMID 31191616
- [Result] Laugel-Haushalter V, Morkmued S, Stoetzel C, Geoffroy V, Muller J, Boland A, Deleuze JF, Chennen K, Pitiphat W, Dollfus H, Niederreither K, Bloch-Zupan A, Pungchanchaikul P. Genetic Evidence Supporting the Role of the Calcium Channel, CACNA1S, in Tooth Cusp and Root Patterning. Front Physiol. 2018 Sep 26;9:1329. doi: 10.3389/fphys.2018.01329. eCollection 2018. PMID 30319441
- [Result] Tardieu C, Jung S, Niederreither K, Prasad M, Hadj-Rabia S, Philip N, Mallet A, Consolino E, Sfeir E, Noueiri B, Chassaing N, Dollfus H, Maniere MC, Bloch-Zupan A, Clauss F. Dental and extra-oral clinical features in 41 patients with WNT10A gene mutations: A multicentric genotype-phenotype study. Clin Genet. 2017 Nov;92(5):477-486. doi: 10.1111/cge.12972. Epub 2017 Mar 19. PMID 28105635
- [Result] Prasad MK, Laouina S, El Alloussi M, Dollfus H, Bloch-Zupan A. Amelogenesis Imperfecta: 1 Family, 2 Phenotypes, and 2 Mutated Genes. J Dent Res. 2016 Dec;95(13):1457-1463. doi: 10.1177/0022034516663200. Epub 2016 Aug 24. PMID 27558265
- [Result] Schossig A, Bloch-Zupan A, Lussi A, Wolf NI, Raskin S, Cohen M, Giuliano F, Jurgens J, Krabichler B, Koolen DA, de Macena Sobreira NL, Maurer E, Muller-Bolla M, Penzien J, Zschocke J, Kapferer-Seebacher I. SLC13A5 is the second gene associated with Kohlschutter-Tonz syndrome. J Med Genet. 2017 Jan;54(1):54-62. doi: 10.1136/jmedgenet-2016-103988. Epub 2016 Sep 6. PMID 27600704
- [Result] Morkmued S, Clauss F, Schuhbaur B, Fraulob V, Mathieu E, Hemmerle J, Clevers H, Koo BK, Dolle P, Bloch-Zupan A, Niederreither K. Deficiency of the SMOC2 matricellular protein impairs bone healing and produces age-dependent bone loss. Sci Rep. 2020 Sep 9;10(1):14817. doi: 10.1038/s41598-020-71749-6. PMID 32908163
- [Derived] Bloch-Zupan A, Rey T, Jimenez-Armijo A, Kawczynski M, Kharouf N; O-Rare consortium; Dure-Molla M, Noirrit E, Hernandez M, Joseph-Beaudin C, Lopez S, Tardieu C, Thivichon-Prince B; ERN Cranio Consortium; Dostalova T, Macek M Jr; International Consortium; Alloussi ME, Qebibo L, Morkmued S, Pungchanchaikul P, Orellana BU, Maniere MC, Gerard B, Bugueno IM, Laugel-Haushalter V. Amelogenesis imperfecta: Next-generation sequencing sheds light on Witkop's classification. Front Physiol. 2023 May 9;14:1130175. doi: 10.3389/fphys.2023.1130175. eCollection 2023. PMID 37228816
- [Derived] Bloch-Zupan A, Huckert M, Stoetzel C, Meyer J, Geoffroy V, Razafindrakoto RW, Ralison SN, Randrianaivo JC, Ralison G, Andriamasinoro RO, Ramanampamaharana RH, Randrianazary SE, Richard B, Gorry P, Maniere MC, Rakoto Alson S, Dollfus H. Detection of a Novel DSPP Mutation by NGS in a Population Isolate in Madagascar. Front Physiol. 2016 Mar 2;7:70. doi: 10.3389/fphys.2016.00070. eCollection 2016. PMID 26973538
- [Derived] Prasad MK, Geoffroy V, Vicaire S, Jost B, Dumas M, Le Gras S, Switala M, Gasse B, Laugel-Haushalter V, Paschaki M, Leheup B, Droz D, Dalstein A, Loing A, Grollemund B, Muller-Bolla M, Lopez-Cazaux S, Minoux M, Jung S, Obry F, Vogt V, Davideau JL, Davit-Beal T, Kaiser AS, Moog U, Richard B, Morrier JJ, Duprez JP, Odent S, Bailleul-Forestier I, Rousset MM, Merametdijan L, Toutain A, Joseph C, Giuliano F, Dahlet JC, Courval A, El Alloussi M, Laouina S, Soskin S, Guffon N, Dieux A, Doray B, Feierabend S, Ginglinger E, Fournier B, de la Dure Molla M, Alembik Y, Tardieu C, Clauss F, Berdal A, Stoetzel C, Maniere MC, Dollfus H, Bloch-Zupan A. A targeted next-generation sequencing assay for the molecular diagnosis of genetic disorders with orodental involvement. J Med Genet. 2016 Feb;53(2):98-110. doi: 10.1136/jmedgenet-2015-103302. Epub 2015 Oct 26. PMID 26502894